CLINICAL TRIAL: NCT02331069
Title: Delto-Tricipital Compression Syndrome: A Randomized Treatment Comparison Trial of Dextrose Injection Versus Physical Therapy.
Brief Title: Delto-Tricipital Compression Syndrome: Treated With Injection of Dextrose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Abierta Interamericana (Other)
Responsible Party: Principal Investigator, Miguel Slullitel, Professor of Orthopedic Surgery, Universidad Abierta Interamericana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAI Protocol number 01006
Record Dates: First submitted 2014-12-17; First posted 2015-01-05 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Superficial Radial Nerve Lesion
Keywords: radial neuropathy
MeSH Terms: conditions — Radial Neuropathy | interventions — Glucose; Water; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dextrose 5% (D5W) Injection (Active Comparator): Glucose injection in 5% concentration, administered weekly X 4 times in a volume of 12 ml or less.
  Interventions: Drug: Dextrose 5% (D5W)
- Physical Therapy (Active Comparator): Physical therapy for a month in the posterior deltoid region 3 times a week.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Drug: Dextrose 5% (D5W) — 0,1,2, and 3 week injection sessions consisting of injection of 2 ml of D5W into the D-T groove at the point of maximal pain at 1-2 cm depth, followed by subcutaneous injection of D5W at 4 cm intervals along the course of the PACN if tenderness is present.
  Other Names: glucose 5% in water
  Arms: Dextrose 5% (D5W) Injection
Other: Physical therapy — Three times weekly X 3 week sessions to include myofascial release, exercise, and one modality.
  Arms: Physical Therapy

SUMMARY:
The posterior antebrachial cutaneous nerve (PACN) can be compressed between the deltoid and triceps, with resultant pain and dysfunction. The active treatment for this study will be injection of the point of compression and along the painful course of the sensory nerve with 5% dextrose. The control treatment will be physical therapy.

DETAILED DESCRIPTION:
The PACN is a purely sensory nerve that originates in the midforearm, courses anterior to the lateral epicondyle, and travels proximally until it dives between the posterior portion of the V shaped insertion of the deltoid and the external? insertion of the triceps, whereupon it joins with the radial nerve.

A proposed pathological explanation is that repetitive co-contraction produces irritation and compression of the nerve at the delto-tricipital (D-T) fascial penetration point. Clinically the patient experiences pain localized to that compression point, and traveling distally along the course of some or all of the posterior femoral cutaneous nerve.

Perineural injection of dextrose has been previously reported for therapeutic use in chronic pain associated with Achilles tendinopathy. Empirically,injection of D5W with a small needle along the course of the PACN and at the D-T penetrator has been found to resolve both pain and dysfunction (describe dysfunction).

Participants will be randomly assigned to either 1 month of physical therapy or to 0,1,2 and 3 week injection of D5W. The use of standardized measurement tools for pain (0-10 numerical rating scale) and function (Quick DASH) will be utilized to determine baseline status and status at 1 month. At 1 month, subjects receiving therapy will be allowed to cross over to injection treatment and all participants will receive as needed treatment until the 1 year period of follow-up. Thus only 1 month data is randomized but long term data will be gathered.

ELIGIBILITY:
Inclusion Criteria:

1. Pain in the deltotricipital groove,extending down the lateral septum.
2. Pain rating 6 or more on a 0-10 numerical rating scale (NRS)
3. Reproduction of pain with provocative maneuvers. Lifting a 6 pound weight to 60 degrees with the below at 40 degrees of elbow extension and the clinician creating a flexion force on the elbow which the participant resists. (Need a picture)
4. Pain more than 3 months?

Exclusion Criteria:

1. Pain in other arm or shoulder locations on either side more than 2/10
2. Pain in other part of the body more than 4/10.
3. Taking narcotics for pain.
4. Pain with testing of shoulder laxity.
5. Massive rupture of rotator cuff (complete width tear) evidenced by examination or MRI scan.
6. Level III-IV or more shoulder arthritis on plain film of shoulder.
7. Other peripheral neuropathy.
8. Unstable psychiatric status

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
NRS Pain (0-10 Numerical Rating Scale) | Time 0 and 1 month
  0-10 Numerical Rating Scale for pain.

SECONDARY OUTCOMES:
Quick Dash Score | Time 0 and 1 month
  Validated shortened version of Disabilities of Arm Shoulder and Hand score.

CONTACTS AND LOCATIONS:
Overall Officials: Mailand Ezequiel, MD, Study Director — Non affiliated; Dean Reeves, Study Chair — Non Affiliated; David Rabago, Study Chair — Non affiliated
Locations (2):
- Argentina (2):
  - Clinica Scanner, Rosario, Santa Fe Province
  - Instituto Jaime Slullitel, Rosario, Santa Fe Province

REFERENCES:
- [Background] Sorensen AA, Howard D, Tan WH, Ketchersid J, Calfee RP. Minimal clinically important differences of 3 patient-rated outcomes instruments. J Hand Surg Am. 2013 Apr;38(4):641-9. doi: 10.1016/j.jhsa.2012.12.032. Epub 2013 Mar 6. PMID 23481405
- [Result] Rabago D, Kijowski R, Woods M, Patterson JJ, Mundt M, Zgierska A, Grettie J, Lyftogt J, Fortney L. Association between disease-specific quality of life and magnetic resonance imaging outcomes in a clinical trial of prolotherapy for knee osteoarthritis. Arch Phys Med Rehabil. 2013 Nov;94(11):2075-82. doi: 10.1016/j.apmr.2013.06.025. Epub 2013 Jul 10. PMID 23850615
- [Result] Yelland MJ, Sweeting KR, Lyftogt JA, Ng SK, Scuffham PA, Evans KA. Prolotherapy injections and eccentric loading exercises for painful Achilles tendinosis: a randomised trial. Br J Sports Med. 2011 Apr;45(5):421-8. doi: 10.1136/bjsm.2009.057968. Epub 2009 Jun 22. PMID 19549615